CLINICAL TRIAL: NCT04348279
Title: Propylene Mesh VS Standard Customized Palatal Stent as Protective Mechanical Barrier Following Harvesting of a Free Palatal Graft: A Short-term Pragmatic Randomized Clinical Trial (Part 1)
Brief Title: Propylene Mesh VS Standard Customized Palatal Stent as Protective Mechanical Barrier
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, PhD holder, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1006
Record Dates: First submitted 2020-04-03; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Randomized Controlled Trial, Human Study
Keywords: palatal wound, propylene mesh, palatal protection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- custom made acrylic stent (Active Comparator): the donor sites of the participants were covered with custom made acrylic stent
  Interventions: Device: propylene mesh
- propylene mesh (Experimental): in the test group, the donor sites received propylene mesh.
  Interventions: Device: propylene mesh

INTERVENTIONS:
Device: propylene mesh — propylene mesh as a palatal stent for palatal wound

SUMMARY:
protection of the palatal wound is an essential step following harvesting a palatal soft tissue graft. During the last decades, several materials were used to avoid protect against the post-operative problems as bleeding, pain and possible infections. The aim of this randomized clinical trial was to assess the usage of polypropylene mesh, compared to the conventional custom-made acrylic stent for efficacy in protection of the palatal wound and reducing the bleeding tendency and post-operative pain. propylene mesh is a promising material for protection of the palatal wound due to its light weight, limited bacterial wicking, tissue compatible properties, however, the custom made acrylic palatal stent provides a more precise mechanical . More studies are required to deeply assess the benefits of this material in the periodontal plastic surgeries.

DETAILED DESCRIPTION:
Background: protection of the palatal wound is an essential step following harvesting a palatal soft tissue graft. During the last decades, several materials were used to avoid protect against the post-operative problems as bleeding, pain and possible infections. The aim of this randomized clinical trial was to assess the usage of polypropylene mesh, compared to the conventional custom-made acrylic stent for efficacy in protection of the palatal wound and reducing the bleeding tendency and post-operative pain.

Patients and methods: A single blinded, parallel group randomized controlled trial took place. Twenty sites were approved to be treated using soft tissue grafting technique with the need for a palatally harvested free graft. The palatal wounds were protected with propylene mesh and custom-made acrylic palatal sten. Participants were qualitatively assessed for bleeding duration, bleeding amount, pain duration, infection possibility, inflammation at 2, 4, 6, 8, 14 days post-operatively. The patient acceptance was also evaluated.

ELIGIBILITY:
Inclusion Criteria:medically free, above 18 years old, non-smokers with healthy reduced periodontium (free of any active disease either gingivitis or periodontitis) -

Exclusion Criteria:During selection, smokers, medically compromised, pregnant and lactating mothers, patients with gagging reflex, incompliant patients, presence of periodontal disease, presence of fixed orthodontic palatal appliance were excluded

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-05-08 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Bleeding intensity | 14 days
  Evaluation of the bleeding amount using VAS test (descriptive tool)
Bleeding duration | 14 days
  Evaluation of the duration of bleeding
Pain level: VAS | 14 days
  evaluation of the pain severity using VAS test (descriptive tool)
pain duration | 14 days
  evaluation of the pain duration

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
if the polypropylene mesh could be used as a palatal protector for the palatal wound following harvesting of a soft tissue graft

REFERENCES:
- [Derived] Yussif N, Wagih R, Selim K. Propylene mesh versus acrylic resin stent for palatal wound protection following free gingival graft harvesting: a short-term pilot randomized clinical trial. BMC Oral Health. 2021 Apr 26;21(1):208. doi: 10.1186/s12903-021-01541-z. PMID 33902550